CLINICAL TRIAL: NCT04439019
Title: Group Education and Digitally Delivered Lifestyle Modification Program to Enable Weight Loss and Improve Metabolic Health and Quality of Life for Patients with Osteoarthritis and Overweight/obesity.
Brief Title: Group Education & Lifestyle Modification's Impact on Weight Loss & Quality Life of Patients with OA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator decision to withdraw study.
Sponsor: Alberta Hip and Knee Clinic (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Kelly Johnston, Assistant Clinical Professor, Alberta Hip and Knee Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB19-1814
Record Dates: First submitted 2020-02-27; First posted 2020-06-19 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Osteo Arthritis Knee; Osteoarthritis, Hip
Keywords: Obesity; carbohydrate restriction; Osteoarthritis; weight loss
MeSH Terms: conditions — Obesity; Osteoarthritis, Hip; Osteoarthritis; Weight Loss

STUDY DESIGN:
Intervention Model Description: The "OA Optimization Program" is a lifestyle and dietary modification program. All Patients will be offered this optional program while they await orthopedic consultation. There is an initial group information session for participants followed by medical assessment which includes medical history and physical examination, a previous dietary history, a readiness for change assessment, and screening for contraindications to the program. The patients will then attend group counselling sessions every 3 months for 1 year, or until their surgical date Patients are encouraged to attend sessions with a family members. We intend to demonstrate improvement in Quality of Life measures including pain and disability in patients with severe osteoarthritis, as well as improvements in markers of health such as BMI, waist circumference, blood pressure, medication use in diabetic and hypertensive patients, and markers such as serum lipids and markers of inflammation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients referred to the Alberta Hip and Knee Clinic (Experimental): All patients who are diagnosed with severe osteoarthritis undergoing total hip/knee replacement surgery and show interest to be part of the study.
  Interventions: Other: Lifestyle and dietary modification program

INTERVENTIONS:
Other: Lifestyle and dietary modification program — The "OA Optimization Program" is a lifestyle and dietary modification program. All Patients will be offered this optional program while they await orthopedic consultation. There is an initial group information session for participants followed by medical assessment which includes medical history and physical examination, a previous dietary history, a readiness for change assessment, and screening for contraindications to the program. The patients will then attend group counselling sessions every 3 months for 1 year, or until their surgical date.Patients are encouraged to attend sessions with a family member. Improvement in Quality of Life measures including pain and disability in patients with severe osteoarthritis, as well as improvements in markers of health such as BMI, waist circumference, blood pressure, medication use in diabetic and hypertensive patients, and markers such as serum lipids and markers of inflammation will be shown.
  Other Names: Osteoarthritis(OA) Optimization program

SUMMARY:
Patients referred to Calgary's Alberta Hip & Knee Clinic, while awaiting consultation with an orthopedic surgeon for hip or knee osteoarthritis, will be offered the opportunity to participate in a dietary counseling program with the goal of attaining weight loss prior to surgery. Those patients interested in participating in the program will be offered the opportunity to participate in the research trial.

DETAILED DESCRIPTION:
Obesity, osteoarthritis, and metabolic syndrome are interrelated diseases. In addition to surgical management, there is the need to identify and provide earlier non-surgical management for individuals with metabolic and body composition changes that are contributing to osteoarthritis progression.

It has been well-established that is a challenge for clinicians to identify and deliver optimal treatment approaches for patients with osteoarthritis and obesity. The long wait times for orthopedic consultation in Alberta present an excellent opportunity to optimize patients with medical comorbidities and can simultaneously improve the pain and disability from their osteoarthritis. This is also an excellent opportunity to involve patients and their families in co-managing their own disease and working towards better health and less pain and disability.

The "OA Optimization Program" has been developed by Dr Berchuk, FRCPC, Diplomat of the American Board of Obesity Medicine. It is a lifestyle and dietary modification program. In cooperation with Calgary's Alberta Hip and Knee Clinic at Gulf Canada Square, Dr Berchuk will offer patients this program while they await orthopedic consultation. This is an optional program offered to all patients. There is an initial group information session for patients who express interest. For those who choose to enroll, the program begins with a medical assessment by Dr Berchuk. The initial consultation consists of a medical assessment which includes medical history and physical examination, a previous dietary history, a readiness for change assessment, and screening for contraindications to the program. The patients will then attend group counselling sessions every 3 months for one year, or until their surgical date. The group counselling will be supplemented by the Grohealth digital therapeutic nutrition program. Participants return for group counselling sessions at Gulf Canada Square clinic every 3 months until orthopedic consultation and if surgery is deemed appropriate, until surgery.

As with any major lifestyle change, peer support is crucial to long term success. Patients are encouraged to bring their family members to the initial consultation and to group sessions. During the group sessions, Dr Berchuk will use techniques to encourage the building of a peer support network, as well as medical cognitive behavior therapy techniques.

Investigators intend to demonstrate that the use of the OA Optimization program can lead to improvement in Quality of Life measures including pain and disability in patients with severe osteoarthritis, as well as improvements in markers of health such as BMI, waist circumference, blood pressure, medication use in diabetic and hypertensive patients, and markers such as serum lipids and markers of inflammation. It is entirely plausible that with preoperative weight loss and/or improvement in metabolic disease, patients may see such dramatic improvement in their symptoms that they choose to postpone surgery.

Research Question and Objectives:

Can the OA Optimization Program lead to improvement in pain and disability related to severe osteoarthritis? Investigators aim to demonstrate that the use of a lifestyle and dietary counselling program can lead to improvements in pain and disability in patients with severe osteoarthritis.

Can the OA Optimization Program demonstrate significant improvements in obesity, hypertension, hyperlipidemia, and glycemic control? Investigators aim to demonstrate improvements in markers of health such as decreased BMI, decreased waist circumference, decreased medication use in diabetic and hypertensive patients, improvement in biomarkers such as serum lipids and serum markers of systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis
* BMI ≥ 25

Exclusion Criteria:

* Age < 18
* Currently following a specialized or therapeutic diet
* Pregnant or breastfeeding
* Type 1 Diabetes
* Unable to read or speak English
* Unwilling to use the digital application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
BMI | every 3 months over 12 months.
  Change in BMI compared to last visit

SECONDARY OUTCOMES:
Blood pressure | every 3 months over 12 months.
  Change in blood pressure compared to last visit
serum lipids and markers of inflammation/ Glycemic acid | every 3 months over 12 months.
  Change in blood markers compared to last visit
Health-related quality of life | every 3 months over 12 months.
  Health-related quality of life as measured by EQ-5D-5L
Pain and functional limitation | every 3 months over 12 months.
  Pain and functional limitation as measured by WOMAC
Medication use | every 3 months over 12 months.
  Changes in use of diabetic and blood pressure medication
waist circumference | every 3 months over 12 months.
  Comparing waist circumference to last visit

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Hip and Knee Clinic, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No